CLINICAL TRIAL: NCT00674687
Title: A Randomized Double-Blind, Placebo-Controlled, Crossover Study To Assess The Reproducibility And The Effect Of Gabapentin On Quantitative Sensory Testing In Neuropathic Pain Patients
Brief Title: A Study Of The Efficacy Of Gabapentin In Neuropathic Pain Patients As Measured By Quantitative Sensory Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A9451138
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-05

CONDITIONS: Neuralgia; Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia; Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Placebo Comparator)
  Interventions: Drug: 2-weeks placebo then gabapentin
- Sequence 2 (Experimental)
  Interventions: Drug: 1-week placebo then gabapentin

INTERVENTIONS:
Drug: 2-weeks placebo then gabapentin — Placebo for 2 weeks followed by gabapentin 300 mg oral capsule once daily titrated over 1 week to gabapentin 600 mg three times daily for 1 week
  Arms: Sequence 1
Drug: 1-week placebo then gabapentin — Placebo for 1 week followed by gabapentin 300 mg oral capsule once daily titrated over 1 week to gabapentin 600 mg three times daily for 2 weeks
  Arms: Sequence 2

SUMMARY:
The purpose of this study is to assess the reproducibility and the effect of gabapentin on quantitative sensory testing assessments in neuropathic pain subjects.

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic pain of peripheral origin as a consequence of either post-herpetic neuralgia or post-traumatic neuropathic pain
* Well-defined skin area of mechanical allodynia to punctate (von Frey filament) stimuli
* Pain intensity score of ≥ 4/10 for von Frey filament-evoked allodynia at the skin area

Exclusion Criteria:

* Patients who have undergone neurolytic or neurosurgical therapy, including skin excisions, for neuropathic pain
* Patients who have trigeminal neuralgia, central pain, chronic radiculopathy, or peripheral neuropathy of non-mechanical or unknown origin
* Patients with any other co-existing pain which cannot be differentiated from the neuropathic pain of peripheral origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Presence/intensity of punctate allodynia (von Frey filament), measured on the pain numeric rating scale (NRS) | Weeks 2 and 4

SECONDARY OUTCOMES:
Subject assessed quality of evoked pain for punctate allodynia | Weeks 2 and 4
Pain NRS score for temporal summation to dynamic brush allodynia (soft and coarse brush) | Weeks 2 and 4
Pressure pain tolerance threshold | Weeks 2 and 4
Pain NRS scores for pressure pain | Weeks 2 and 4
Subject assessed quality of evoked pain for temporal summation to dynamic brush allodynia (soft and coarse brush) | Weeks 2 and 4
Tactile threshold | Week 4
Pressure pain detection threshold | Weeks 2 and 4
Area of punctate and dynamic (soft and coarse brush) allodynia | Weeks 2 and 4
Pain NRS score for punctate allodynia | Weeks 2 and 4
Pain NRS scores for temporal summation to punctate stimuli | Weeks 2 and 4
Subject assessed quality of evoked pain for temporal summation to punctate stimuli | Weeks 2 and 4
Neuropathic pain scale | Week 4
Test-day global pain scale | Week 4
Pain diary card | Week 4
Pain NRS score for dynamic brush allodynia (soft brush) | Weeks 2 and 4
Subject assessed quality of evoked pain for dynamic brush allodynia (soft brush) | Weeks 2 and 4
Presence of metabonomic biomarkers | Weeks 1 and 4
Physical examination | 1 week after 4-week treatment period
Adverse events | Throughout study duration
Clinical laboratory tests | 1 week after 4-week treatment period
Subject assessed quality of pressure pain | Weeks 2 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Liverpool, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451138&StudyName=A%20Study%20Of%20The%20Efficacy%20Of%20Gabapentin%20In%20Neuropathic%20Pain%20Patients%20As%20Measured%20By%20Quantitative%20Sensory%20Testing